CLINICAL TRIAL: NCT04807673
Title: A Multicenter Randomized, Controlled Phase III Clinical Trial of Pembrolizumab Plus Paclitaxel and Cisplatin Versus Neoadjuvant Chemoradiotherapy Followed by Surgery for Locally Advanced Esophageal Squamous Cell Carcinoma (KEYSTONE-002)
Brief Title: Pembrolizumab Plus Neoadjuvant Chemotherapy vs. Neoadjuvant Chemoradiotherapy for Locally Advanced ESCC (KEYSTONE-002)
Acronym: KEYSTONE-002
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Shanghai Chest Hospital (Other); Ruijin Hospital (Other); Hebei Medical University Fourth Hospital (Other); Harbin Medical University (Other); Liaoning Cancer Hospital & Institute (Other); Shanxi Province Cancer Hospital (Other); Jining First People's Hospital (Other); Weifang People's Hospital (Other); Tianjin Medical University General Hospital (Other); Shandong Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TianjinCIH20210096
Record Dates: First submitted 2021-03-11; First posted 2021-03-19 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; Immunotherapy; neoadjuvant therapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — pembrolizumab; Paclitaxel; Cisplatin; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab+ Paclitaxel+Cisplatin+ Surgery+Pembrolizumab (228) (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 every 3 weeks (Q3W), paclitaxel 135mg/m^2 IV on Day 2 Q3W, and cisplatin 80 mg/m^2 IV on Day 2 Q3W, a total of three cycles. All treatments will be beginning on Day 1 of each 3-week dosing cycle. Surgery should be done within 4-6 weeks after the last neoadjuvant treatment. After surgery, pembrolizumab 200 mg IV on Day 1 Q3W lasting one year.
  Surgery: McKeown esophagectomy
  Interventions: Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Cisplatin
- neoadjuvant chemoradiotherapy+ Surgery (114) (Experimental): neoadjuvant chemoradiotherapy 41.4Gy(1.8Gy×23 fractions) with five cycles of TP(Paclitaxel 50mg/m^2 on D1 and Cisplatin 25mg/m^2 D1, repeated every week. Surgery should be done within 4-6 weeks after the last neoadjuvant treatment.
  Surgery: McKeown esophagectomy
  Interventions: Radiation: neoadjuvant chemoradiotherapy

INTERVENTIONS:
Biological: Pembrolizumab — Neoadjuvant period: pembrolizumab 200mg IV D1, Q3W, and preoperative therapy with three cycles.
  Adjuvant period: pembrolizumab 200 mg IV D1, Q3W, up to one year, which should be performed within 3-6 weeks after surgery.
  Other Names: Keytruda
  Arms: Pembrolizumab+ Paclitaxel+Cisplatin+ Surgery+Pembrolizumab (228)
Drug: Paclitaxel — Neoadjuvant period: paclitaxel 135mg/m^2 IV on Day 2 Q3W, and a total of three cycles.
  Arms: Pembrolizumab+ Paclitaxel+Cisplatin+ Surgery+Pembrolizumab (228)
Drug: Cisplatin — Neoadjuvant period: cisplatin 80 mg/m^2 IV on Day 2 Q3W, and a total of three cycles.
  Arms: Pembrolizumab+ Paclitaxel+Cisplatin+ Surgery+Pembrolizumab (228)
Radiation: neoadjuvant chemoradiotherapy — neoadjuvant chemoradiotherapy 41.4Gy(1.8Gy×23 fractions) with five cycles of TP(Paclitaxel 50mg/m^2 on D1 and Cisplatin 25mg/m^2 D1, repeated every week
  Arms: neoadjuvant chemoradiotherapy+ Surgery (114)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pembrolizumab plus paclitaxel, cisplatin as neoadjuvant therapy followed by surgery, and pembrolizumab as adjuvant therapy, compared with neoadjuvant chemoradiotherapy and surgery for locally advanced ESCC in multicenter.

DETAILED DESCRIPTION:
Preoperative chemoradiotherapy with radical surgery is the recommended treatment for locally advanced esophageal squamous cell carcinoma (ESCC) in the NCCN guidelines. But many patients refused or abandon radiotherapy because of the intolerable adverse effects. The purpose of this study is to evaluate the efficacy and safety of pembrolizumab plus paclitaxel, cisplatin as neoadjuvant therapy followed by surgery, and pembrolizumab as adjuvant therapy, compared with neoadjuvant chemoradiotherapy and surgery for locally advanced ESCC in multicenter. The primary study hypothesis is that Event Free Survival (EFS) is superior with pembrolizumab plus neoadjuvant chemotherapy compared with neoadjuvant chemoradiotherapy in participants with ESCC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed esophageal squamous cell carcinoma;
2. R0 resectable thoracic esophageal cancer, cT1-3N1-2M0, cT2-3N0M0 (AJCC V8 TNM classification);
3. No suspicious metastatic lymph nodes on the clavicle;
4. Have a performance status of 0 or 1 on the ECOG Performance Scale;
5. Age 18-75 years old, both men and women;
6. Be willing and able to provide written informed consent/assent for the trial;
7. Demonstrate adequate organ function ;
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours before receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required;
9. Be willing to provide tissue, blood, and urine samples. Tissue should be from a newly obtained core or excisional biopsy of a tumor lesion through repeated biopsies. Newly-obtained is defined as a specimen obtained up to 4 weeks (28 days) before initiation of treatment on Day 1.
10. Have not received systemic or local treatment for esophageal cancer in the past.

Exclusion Criteria:

1. Ineligibility or contraindication for esophagectomy;
2. Prior therapy (operation, radiotherapy, immunotherapy, or chemotherapy) for esophageal cancer
3. Active autoimmune disease or history of autoimmune disease;
4. Requiring systemic treatment with either corticosteroids or other immunosuppressive medications;
5. Subjects with a history of symptomatic interstitial lung disease;
6. History of allergy to study drug components;
7. Women must not be pregnant or breast-feeding;
8. Patient has received prior chemotherapy, radiotherapy, target therapy ，and immune therapy for this malignancy or any other past malignancy;
9. Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | Up to approximately 2.5 years
  EFS is defined as the time from randomization to the first documented disease progression per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by investigator, or recurrence, or metastasis, or death due to any cause, whichever occurs first. For this analysis, EFS will be assessed in participants with ESCC.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 and 5 years
  OS is defined as the time from randomization to death due to any cause.
Disease Free Survival (DFS) | 3 and 5 years
  Percentage of Participants With DFS, as Assessed by RECIST 1.1. DFS is defined as the time from randomization to the first documented disease progression of local recurrence or distant metastasis or death due to any cause.
Major pathologic response (MPR) | 1 month after resection
  MPR is defined as viable tumor comprised ≤ 10% of resected tumor specimens.
Objective response rate (ORR) | 1 month after resection
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by investigator. For this analysis, ORR will be assessed in all participants.
Pathologic Complete Response (PCR) | 1 month after resection
  PCR is defined as pT0N0M0
assessment in perioperation | perioperative period
  R0 resection rate， Time of operation， Quantity of bleeding， Thoracic Drainage， Days of Hospitalization， Rate of Operative Complication， Mortality of perioperation
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 16 months
  All participants with treatment-related adverse events as assessed by National Cancer Institute Common Terminology Criteria for Adverse Event,Version 4.0(CTC AE4.0).
Quality of life differences (EORTC QLQ-C30) | 2.5 years
  The quality of life will be assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer patients (EORTC QLQ-C30) questionnaire. Patients will be invited to finish the questionnaire at the first day of randomization, before surgery and after surgery (3m, 6m, 12m and 24 months).
Quality of life differences (EORTC QLQ-OES18) | 2.5 years
  The quality of life will be assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer patients (EORTC QLQ-OES18) questionnaire. Patients will be invited to finish the questionnaire at the first day of randomization, before surgery and after surgery (3m, 6m, 12m and 24 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of minimally invasive esophageal surgery, Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Batran SE, Koch C. Neoadjuvant therapy for oesophageal cancer: refining the armamentarium. Lancet. 2024 Jul 6;404(10447):5-7. doi: 10.1016/S0140-6736(24)01084-5. Epub 2024 Jun 11. No abstract available. PMID 38876135
- [Derived] Shang X, Zhang W, Zhao G, Liang F, Zhang C, Yue J, Duan X, Ma Z, Chen C, Pang Q, Zhang W, Liu L, Ren X, Meng B, Zhang P, Ma Y, Zhang L, Li H, Kang X, Li Y, Jiang H. Pembrolizumab Combined With Neoadjuvant Chemotherapy Versus Neoadjuvant Chemoradiotherapy Followed by Surgery for Locally Advanced Oesophageal Squamous Cell Carcinoma: Protocol for a Multicentre, Prospective, Randomized-Controlled, Phase III Clinical Study (Keystone-002). Front Oncol. 2022 Mar 31;12:831345. doi: 10.3389/fonc.2022.831345. eCollection 2022. PMID 35433421